CLINICAL TRIAL: NCT01563419
Title: Clinical Usefulness of a Magnifier for Insulin Pen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Cho, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: magnifier
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus
Keywords: Insulin; Diabetes; Low vision
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Vision, Low

ARMS (2):
- Control (No Intervention): dialing up the selected dose of insulin pens without an indicator magnifying window
- Magnifier (Experimental): dialing up the selected dose of insulin pens clipped on an indicator magnifying window
  Interventions: Device: Indicator magnifying window (Izumi Planning Co.)

INTERVENTIONS:
Device: Indicator magnifying window (Izumi Planning Co.) — IZUMI PLANNING CO,.LTD.Tokyo.Japan
  Material: Polypropylene with polycarbonate lens
  Arms: Magnifier

SUMMARY:
Insulin treatment is crucial for glucose control. Many patients with type 2 diabetes exhibit inadequate glycemic control in spite of combination of oral antidiabetic drugs and eventually need insulin therapy. Patients who need insulin therapy are older and have poor visual acuity, which predispose to inaccurate dosing and consequent hyper or hypoglycemia.In this study, the investigators examined the clinical usefulness of a magnifier for elderly diabetic patients who had used insulin pens.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes mellitus
* over 60 years old
* who have self-injected insulin with insulin pens

Exclusion Criteria:

* who have visual acuity less than 20/200 for each eye
* who had surgery on his/her eyes within a week

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
the time spent to complete dialing up insulin pens | from to start dialing up the selected dose to to complete dialing up, assessed up to 10 minutes
  The investigators ask participants to dial up the random dose of insulin pens between 30 and 40 and measured the time spent to complete dialing up.

SECONDARY OUTCOMES:
the dosing accuracy | from to start dialing up the selected dose to to complete dialing up, assessed up to 10 minutes
  The investigators ask participants to dial up the random dose of insulin pens between 30 and 40 and check whether they dial up the selected dose correctly.
the convenience in using insulin pens | the duration of to complete filling up the questionnaires, an expected average of 10 minutes
  By structured questionnaires, the investigators ask participants about the convenience in dialing up to correct doses of insulin pens.
the self-confidence in using insulin pens | the duration of to complete filling up the questionnaires, an expected average of 10 minutes
  By structured questionnaires, the investigators ask participants about the self-confidence in dialing up to correct doses of insulin pens
the need for glasses in using insulin pens | the duration of to complete filling up the questionnaires, an expected average of 10 minutes
  By structured questionnaires, the investigators ask participants about the need for glasses in dialing up to correct doses of insulin pens
the preferences for the use of a magnifier | the duration of to complete filling up the questionnaires, an expected average of 10 minutes
  By structured questionnaires, the investigators ask participants whether they prefer the use of a magnifier
the recommendation for the use of a magnifier | the duration of to complete filling up the questionnaires, an expected average of 10 minutes
  By structured questionnaires, the investigators ask participants whether they recommend the use of a magnifier to others.

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD,PhD, Study Chair — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea